CLINICAL TRIAL: NCT06560684
Title: A PHASE 2 CROSSOVER STUDY OF ON-DEMAND PREP FORMULATIONS COMPARING RECTAL AND ORAL TENOFOVIR-BASED PREP EVALUATING EXTENDED SAFETY, ACCEPTABILITY, AND PHARMACOKINETICS/PHARMACODYNAMICS
Brief Title: CROSSOVER STUDY OF ON-DEMAND PREP FORMULATIONS COMPARING RECTAL AND ORAL TENOFOVIR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HPTN 106
Record Dates: First submitted 2024-08-02; First posted 2024-08-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-07

CONDITIONS: Tenofovir
Keywords: PrEP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Those participants assigned to Group A will start with the rectal TFV 660 mg douche for the first 8 weeks (Period 1) and then after a 2-4 week washout will switch to the on-demand oral F/TDF 200 mg/300 mg sequence for the next 8 weeks (Period 2).
  Interventions: Drug: Oral F/TDF Pills; Drug: TFV rectal douche
- Group B (Experimental): Those participants assigned to Group B will start with the on-demand oral F/TDF 200 mg/300 mg sequence for 8 weeks and then after a 2-4 week washout will switch to the rectal TFV 660 mg douche for the next 8 weeks (Period 2).
  Interventions: Drug: Oral F/TDF Pills; Drug: TFV rectal douche

INTERVENTIONS:
Drug: Oral F/TDF Pills — For 8 weeks of each study period, the participant will take the study product at least weekly prior to anticipated RAI.
Drug: TFV rectal douche — For 8 weeks of each study period, the participant will take the study product at least weekly prior to anticipated rectal anal intercourse (RAI).

SUMMARY:
This is a Phase 2, multi-site, two-period, open label randomized crossover (Period 1 and 2) study. Participants are randomized 1:1 to one of two 8-week on-demand product sequences - TFV douche then oral F/TDF or oral F/TDF then TFV douche - with a 2 to 4-week washout period in between. Domains of safety, acceptability, adherence, and PK/PD (sub-study only) are assessed for each product.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 years or older at the time of screening informed consent
2. Willing and able to provide informed consent to take part in the study
3. Able to read at a level required for the study components (e.g., CASI and SMS)
4. Have access to device and the internet for completion of study procedures
5. Understand and agree to local STI reporting requirements
6. Non-reactive/negative HIV test results at screening and enrollment
7. A history of consensual RAI at least five times in their lifetime and at least once in the prior 3 months
8. Received or self-administered an enema or rectal douche more than half the time prior to engaging in RAI in the past year.
9. Willing and able to use condoms for all sexual intercourse for the duration of participation
10. Agrees not to participate in other research studies involving drugs, biologics, medical devices, vaccines, anal products, or genital products for the duration of the study
11. Willing and able to provide adequate locator information
12. Agrees not to knowingly engage in receptive or insertive sexual activity with another study participant for the duration of study participation.
13. Available to return for all study visits and within any site's catchment area

ADDITIONAL INCLUSION FOR THOSE IN THE PK/PD SUB-STUDY

1. Willing to refrain from occasional over-the-counter use of aspirin and NSAID use for 72 hours before and after each study biopsy visit
2. Willing to abstain from insertion of anything (e.g., drug/medication, penis, object, sex toy, or enema including take-home enema) into the anorectum for 72 hours before study drug dose and until 72 hours after each flexible sigmoidoscopy with biopsy collection, or one week after the study drug dose, whichever is later
3. Willing and able to use specific condoms and lubricant provided by the study clinic for all RAI for the duration of participation

Exclusion Criteria:

1. Any reactive/positive HIV test at screening or at least one reactive/positive test result at enrollment, even if HIV infection is not confirmed
2. History of active (including chronic) hepatitis B virus (HBV) infection, as documented by positive HBV surface antigen (HBsAg) at screening
3. Co-enrollment in any other interventional research study that may interfere with this study (as provided by self-report or other available documentation). Exceptions may be made after consultation with the Clinical Management Committee (CMC).
4. ≥ Grade 2 clinically significant laboratory abnormality at baseline as defined by The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017, except for estimated glomerular filtration rate (eGFR), which must be >75 mL/min/1.73m^2. (Coagulation (PT/INR) results ≥ Grade 2 are not exclusionary for the main study).
5. Significant colorectal symptom(s) as determined by medical history or by participant self-report (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, history of inflammatory bowel disease, presence of symptomatic external hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation)
6. At screening, participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current CDC guidelines or symptomatic urinary tract infection (UTI)

   a.Infections requiring treatment include chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts.

   Note: if an STI apart from HIV is detected, the participant will be referred for treatment and, upon documented confirmation of definitive treatment, can be retested in three weeks for evidence of adequate treatment.
7. History of an underlying clinically significant cardiac arrhythmia or renal disease
8. History of severe or recent cardiac or pulmonary event
9. History of significant gastrointestinal bleeding
10. Use of F/TDF or use of F/TAF as HIV PrEP within 8 weeks prior to screening visit or anticipated use throughout study participation
11. Use of injectable PrEP within 8 weeks prior to the screening visit or anticipated use throughout study participation
12. Use of systemic or anorectal immunomodulatory medications, rectally administered products containing N-9 or corticosteroids, or any investigational products unless otherwise permitted within 4 weeks of screening or planned use at any time during study participation
13. Known allergic reaction to TFV or other components of the test articles
14. Current known partners with HIV, unless with sustained viral suppression on antiretroviral treatment (ART)
15. History of recurrent urticaria
16. Symptoms suggestive of acute HIV infection at screening or enrollment
17. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease

ADDITIONAL EXCLUSION FOR THOSE IN THE PK/PD SUB-STUDY

1. Current medically-indicated use of warfarin or heparin or other anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], non-steroidal anti-inflammatory drugs [NSAIDs], or Pradaxa®)
2. Previous use of injectable PrEP
3. ≥ Grade 2 laboratory result for coagulation testing (PT/INR) at baseline as defined by The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Grade 2 or higher adverse events during each study Period | Week 1 through 19
  For eGFR, participants may enroll in the study with an eGFR value consistent with a grade 2 adverse event; thus, an exception will be made for eGFR, which will be considered a safety outcome if it worsens to a grade 3 or higher.
Any adverse event leading to study product discontinuation during each study Period | Week 1 through 19
Self-report on ease of use, product liking, and likelihood of future use during each study Period | Week 1 through 19
  measured via computer-assisted self-interview (CASI), with the scales for the specific questions ranging from 1 (lowest ranking) to 4 (highest ranking).

SECONDARY OUTCOMES:
Proportion of participants who reported being most likely to use the TFV douche in the future (following Period 2) | Week 1 through 19
Percent prescribed weekly doses taken in each Period using multiple subjective and objective measures | Week 1 through 19
TFV and FTC concentrations in blood plasma and rectal tissue biopsies | Week 1 through 19
  (Sub-study only)
TFV-DP and FTC-TP concentrations in PBMCs, rectal tissue biopsies, and mucosal mononuclear cells (MMC) | Week 1 through 19
  (Sub-study only)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Alabama CRS (Site ID# 31788), Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Hope Clinic CRS, Lawrenceville, Georgia
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Weill Cornell Chelsea CRS, New York, New York
  - Chapel Hill CRS (3201), Chapel Hill, North Carolina
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No